CLINICAL TRIAL: NCT02939690
Title: Estimation of Umbilical Venous Catheter Insertion Depth in Newborns Using Weight or Body Measurement: A Randomized Trial
Brief Title: Umbilical Venous Catheter Insertion Depth in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Amuchou Soraisham, Associate Professor of Pediatrics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16-1303
Record Dates: First submitted 2016-09-22; First posted 2016-10-20 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Central Venous Catheterization
Keywords: Catheter; Umbilical vein; Neonate
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UVC and surface measurement formula (Experimental): UVC insertion depth = Umbilicus to nipple distance minus 1cm
  Interventions: Device: UVC; Device: Ultrasound
- UVC and Birth weight based formula (Active Comparator): UVC insertion depth=[(3× birth weight (Kg) + 9)/2+1)] cm
  Interventions: Device: UVC; Device: Ultrasound

INTERVENTIONS:
Device: UVC — UVC insertion depth calculated by [(3× birth weight (Kg) + 9)/2+1)]
  Other Names: UVC insertion using birth weight based calculation
  Arms: UVC and Birth weight based formula
Device: UVC — UVC insertion depth calculated by umbilicus to nipple distance-1
  Other Names: UVC insertion using surface measurement
  Arms: UVC and surface measurement formula
Device: Ultrasound
  Other Names: Ultrasound assessment of UVC

SUMMARY:
In this randomized clinical study, neonates who require umbilical venous catheter (UVC) insertion as part of their routine care at anytime during their NICU admission will be randomized to one of the 2 formulas for estimation of the pre-insertion UVC depth (umbilicus to the nipple in cm minus 1 (UN - 1) or birth weight based formula ([(3× birth weight (Kg) + 9)/2+1)]. UVC will be inserted under sterile condition as per unit protocol. To verify the UVC tip position, a thoracoabdominal radiograph will be taken. In addition, the investigators will do a ultrasound of the heart to assess the exact location of the catheter tips as soon as possible but within 6 hours of insertion.

DETAILED DESCRIPTION:
Background:

The ideal position of UVC) tip to minimize complications is just outside the heart at the junction of inferior vena cava and right atrium. UVC related complications are mainly due to catheter malposition. Accurate prediction of insertion length of UVC as well as confirmation of the position after insertion by radiograph or with ultrasound is very important to avoid complications. UVC malposition with subsequent re-positioning exposes these fragile infants to unnecessary handling, further radiologic exposure and increasing risk of infection.

The commonly used formulas to estimate the depth of umbilical catheter include Dunn's shoulder to umbilical length graph and a birth weight based formula proposed by Shukla and Ferrara in 1986. In Calgary, the most commonly used method for estimation of UVC insertion length is the birth weight based formula (i.e. UVC insertion length = (3 x birth weight + 9)/2 +1). The success rate of achieving the optimum position of catheter tip using this formula ranges from 31-40%. A recent retrospective study reported the use of different surface markers for calculating UVC insertion depth. A distance from base of umbilicus to nipple distance (UN)-1 cm provided the best and most accurate insertion depth of UVC. This formula had accuracy rate of 84% compared with 57% accuracy rate with birth weight based formula.

The objectives of our study are:

1. To compare accuracy rate between UVC insertion length estimated by using two formula (i.e. umbilicus to the nipple distance in cm minus 1 (UN - 1) and Shukla's birth weight based formula ([(3× birth weight (Kg) + 9)/2+1)] in achieving optimum UVC tip position
2. To compare the accuracy rate of UVC tip position between two methods based on growth status of neonates

Methods:

This is a randomized clinical study. All infants who require UVC insertion as part of their routine care at anytime during their hospital admission are eligible for the study. Infants with hydrops fetalis, abdominal wall defects, congenital diaphragmatic hernia and/or major structural heart disease will be excluded from the study.

When a newborn baby needs UVC central line insertion, neonate will be randomized to one of the 2 formulas for estimation of the pre-insertion UVC depth. UVC will be inserted under sterile condition as per unit protocol. To verify the UVC tip position, a thoracoabdominal radiograph will be taken. In addition,the investigators will do a ultrasound of the the heart to assess the exact location of the catheter tips as soon as possible but within 6 hours of insertion.

ELIGIBILITY:
Inclusion Criteria:

* All infants who require UVC insertion as part of their routine care at anytime during their NICU admission

Exclusion Criteria:

* Infants with hydrops fetalis, infants with abdominal wall defects, congenital diaphragmatic hernia and major structural heart disease

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Proportion of correctly inserted UVC at optimum catheter tip position | within 12 hours

SECONDARY OUTCOMES:
Number of readjustment of UVC | within first 2 weeks
Comparison of UVC tip position between two methods based on based growth status at birth (i.e.AGA, SGA, LGA) | within 12 hours
  AGA: appropriate for gestational age (i.e birth weight between 10th and 90th percentile for gestational age); SGA: Small for gestational age (i.e. birth weight <10th percetile for gestational age); LGA: large for gestational age (i.e.birth weight >90th percentile for gestational age) using Fentons growth chart for preterm infants and WHO growth chart for term infants

CONTACTS AND LOCATIONS:
Overall Officials: Amuchou S Soraisham, MD, DM,, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shukla H, Ferrara A. Rapid estimation of insertional length of umbilical catheters in newborns. Am J Dis Child. 1986 Aug;140(8):786-8. doi: 10.1001/archpedi.1986.02140220068034. PMID 3728405
- [Result] Gupta AO, Peesay MR, Ramasethu J. Simple measurements to place umbilical catheters using surface anatomy. J Perinatol. 2015 Jul;35(7):476-80. doi: 10.1038/jp.2014.239. Epub 2015 Jan 22. PMID 25611793
- [Result] Kieran EA, Laffan EE, O'Donnell CP. Estimating umbilical catheter insertion depth in newborns using weight or body measurement: a randomised trial. Arch Dis Child Fetal Neonatal Ed. 2016 Jan;101(1):F10-5. doi: 10.1136/archdischild-2014-307668. Epub 2015 Aug 11. PMID 26265678
- [Result] Harabor A, Soraisham A. Rates of intracardiac umbilical venous catheter placement in neonates. J Ultrasound Med. 2014 Sep;33(9):1557-61. doi: 10.7863/ultra.33.9.1557. PMID 25154935
- [Result] Michel F, Brevaut-Malaty V, Pasquali R, Thomachot L, Vialet R, Hassid S, Nicaise C, Martin C, Panuel M. Comparison of ultrasound and X-ray in determining the position of umbilical venous catheters. Resuscitation. 2012 Jun;83(6):705-9. doi: 10.1016/j.resuscitation.2011.11.026. Epub 2011 Dec 6. PMID 22155219
- [Result] Dunn PM. Localization of the umbilical catheter by post-mortem measurement. Arch Dis Child. 1966 Feb;41(215):69-75. doi: 10.1136/adc.41.215.69. No abstract available. PMID 5906629
- [Derived] Sheta A, Kamaluddeen M, Soraisham AS. Umbilical venous catheter insertion depth estimation using birth weight versus surface measurement formula: a randomized controlled trial. J Perinatol. 2020 Apr;40(4):567-572. doi: 10.1038/s41372-019-0456-0. Epub 2019 Aug 5. PMID 31383945